CLINICAL TRIAL: NCT03941119
Title: VRx: Randomized Controlled Trial to Evaluate the Impact of Virtual Reality Therapy on Behavioural and Psychological Symptoms and Quality of Life of Individuals With Dementia Admitted to an Acute Care Hospital
Brief Title: Evaluating the Impact of VR-therapy on BPSD and QoL of Individuals With Dementia Admitted to Hospital
Acronym: VRx-RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: All recruitment activities for this study (with acutely ill inpatients with dementia) stopped due to the COVID pandemic.
Sponsor: University Health Network, Toronto (Other)
Collaborators: Centre for Aging and Brain Health Innovation (Other); Michael Garron Hospital (Other)
Responsible Party: Principal Investigator, Lora Appel, Collaborating Scientist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 782-1812-Mis-332
Record Dates: First submitted 2019-01-15; First posted 2019-05-07 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Dementia; Delirium Superimposed on Dementia
Keywords: Virtual Reality; Biomedical Technology; Non-pharmacological Intervention; Behavioral Symptoms; Quality of Life; Geriatric Nursing; Health Services for the Aged; Hospitals, Community; Cognitive Dysfunction; Dementia; Delirium
MeSH Terms: conditions — Dementia; Behavioral Symptoms; Cognitive Dysfunction; Delirium

STUDY DESIGN:
Intervention Model Description: This is an open trial, unblinded to both participants and research staff, due to the nature of the intervention. The randomization into VR-therapy or standard of care (no VR-therapy) will be performed using a randomization tool within a secure web application. The sequence allocation will be concealed from those assigning participants to the intervention groups, until the moment of assignment. Participants will be assigned to groups only after informed consent has been obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will receive a VR-therapy session every 24-72 hours of their stay in the hospital. Participants will view specially designed 360-degree VR films using a Virtual Reality head mounted display for a maximum of 20 minutes per session.
  Interventions: Other: VR-therapy
- Control (No Intervention): The control arm will not receive any VR-therapy sessions during their hospital stay.

INTERVENTIONS:
Other: VR-therapy — Wearing a Virtual Reality head mounted device allows the user to become immersed in a virtual environment. We have assembled a library of 3-10 minute 360-degree films from a variety of nature settings. The VR films were intentionally chosen to be calming in distinctive ways, as supported by the literature around nature visualization and wellbeing. By varying 1) the lengths of the films (3, 5, and 10 minutes), 2) the types of natural elements (greenery, earth, sky, water), 3) distance of view (close-ups, vistas), 4) motion (flowing water, wind in trees), 5) sound, and 6) presence of different elements (humans/animals, scenery, urban sites, etc.), the content provides a wide range of attributes that can be collaboratively selected by the individual, caregiver, or health care provider for each individual. We will display these films on commercially available VR equipment and will provide audio matching the film using commercially available headphones.
  Other Names: Oculus Go Standalone Virtual Reality Headset; Oculus Go; Virtual Reality Headset; VR Headset; VR HMD; Virtual Reality
  Arms: Intervention

SUMMARY:
Behavioural and Psychological Symptoms of Dementia (BPSD) (such as aggression, restlessness, agitation, wandering, anxiety, depression) are common to most people with dementia at some point during their illness and represent an aspect of dementia particularly difficult to manage. There is growing attention to the therapeutic effects of natural environments on people's health. Exposure to natural environments (seeing greenery, hearing outside natural sounds) has been shown to enhance wellbeing, reduce depression, anxiety and stress levels, and decrease hospital length-of-stay for inpatients. Virtual Reality (VR) is a novel technology that uses a Head Mounted Display (HMD) to generate simulated immersive experiences that elicit perceptions and behaviors similar to those in real life and can make one feel as though they are truly present in another place. Based on scientific research, previous studies, and expert consultation, we created a library of VR experiences depicting calming nature scenes designed specifically for people with dementia.

The objectives of this RCT are 1) to evaluate the effects of VR-therapy on BPSD and the hospital care experience of in-patients with dementia and/or delirium admitted to an acute care hospital, 2) to determine the usability, tolerability, and safety of VR-therapy for patients with dementia and/or delirium admitted to acute care, 3) determine the effect of VR-therapy on quality of life for patients with dementia and/or delirium admitted to acute care and 4) to explore a framework for introducing non-pharmacological therapies in acute care hospitals.

Our hypotheses are 1) VR-therapy helps manage BPSD (e.g. decrease anxiety, aggression, depression, violent behaviors, incidents of wandering), and may decrease the amount and/or frequency of sedatives and anti-depressant medication administered and/or the number of incidents that require restraints, and the number of falls, in people with dementia and/or delirium admitted to an acute care hospital. 2) VR-therapy will improve the quality of life for individuals with dementia and/or delirium admitted to an acute care hospital (operationalized through conducting a validated instrument to measure quality of life for people with dementia). 3) VR-therapy is safe and feasible to administer to individuals with dementia and/or delirium admitted to an acute care hospital (with assistance from their circle of care members and/or caregivers).

DETAILED DESCRIPTION:
Behavioural and Psychological Symptoms of Dementia (BPSD) (including hallucinations, delusions, aggression, restlessness, agitation, wandering, anxiety, depression, elation, euphoria, disinhibition, motor disturbances, nighttime behaviours, and appetite disturbances) represent an aspect of dementia particularly difficult to manage for which new treatments are urgently needed. Current means to manage BPSD typically involve medications (e.g. anti-psychotics, anti-depressants, sedatives) associated with negative side effects such as lethargy, loss-of-self, cognitive decline, and increased risk of falls, and/or applying physical barriers and restraints (alarms, locks, Buxton chairs, tethers) that can cause pressure sores, injury, infection, as well as negative psychological effects such as anxiety, distress, and aggression. Although options for non-pharmacological management of BPSD in acute care exist (e.g. reminiscence therapy, therapeutic touch, music therapy), they are seldom implemented in practice due to lack of time, resources, and/or training.

Exposure to natural environments (seeing greenery, hearing outside natural sounds) has been shown to enhance wellbeing, reduce depression, anxiety, and stress levels, and decrease hospital length-of-stay for inpatients. Through VR technology, one's surroundings can be seamlessly replaced by a virtual world of their choosing. Based on previous studies and expert consultation, we created a library of VR experiences depicting calming nature scenes (peaceful lake, refreshing forest, cheerful playground) designed specifically for people with dementia, as a prototype for introducing immersive VR-therapy to hospitals, long term care facilities and private homes. The goal of VR-therapy is to help manage BPSD and stimulate psychological/cognitive health and daytime engagement for people with dementia.

The RCT will be informed by our prior pilot study conducted in the hospitalist medicine department of Michael Garron Hospital with inpatients with dementia to validate the proposed RCT study protocol (processes, methods, recruitment strategy, resource requirements, timelines) as well as by previous feasibility studies in outpatients that showed it is safe and feasible to use VR/HMDs for people with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 65 years of age or older.
* Patients admitted to Michael Garron Hospital (MGH).
* Patients diagnosed with, or suspected to have, dementia.

Exclusion Criteria:

* Patients with open wounds on face (sutured lacerations exempted).
* Patients with a history of seizures or epilepsy.
* Patients with a pacemaker.
* Patients with head trauma or stroke leading to their current admission.
* Patients with cervical conditions or injuries that would make it unsafe for them to use the VR headset.
* Patients with alcohol related dementia/ Korsakoff syndrome.
* Patients admitted to the Intensive Care Unit (ICU) or Adult Mental Health Inpatient Service.
* Patients who require but do not have a Substitute Decision Maker (SDM) or patients from which there is no contactable SDM.
* Patients who have a Public Guardian and Trustee (PGT) as SDM.
* Patients who participated in the VRx study during their previous hospitalization and are readmitted less than 30-days after previous hospital discharge.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Changes in Behavioural and Psychological Symptoms of Dementia (BPSD) during the hospital stay | Throughout the acute hospitalization, an average of 10.6 days
  BPSD recorded in the electronic medical record during the acute hospitalization, averaging 10.6 days, will be assessed for all participants. The E-BEHAVE-AD will be administered to all participants on days 1 and 4-7 of hospitalization
Number of falls without injury during the hospital stay | Throughout the acute hospitalization, an average of 10.6 days
  All falls without injury that occurred during the current acute hospitalization that were recorded in the electronic medical record will be assessed for all participants
Number of falls with injury during the hospital stay | Throughout the acute hospitalization, an average of 10.6 days
  All falls with injury that occurred during the acute hospitalization that were recorded in the electronic medical record will be assessed for all participants
Number of pressure ulcers during the hospital stay | Throughout the acute hospitalization, an average of 10.6 days
  All pressure ulcers that developed during the acute hospitalization that were recorded in the electronic medical record will be assessed for all participants
All-cause in-patient mortality during the hospital stay | Throughout the acute hospitalization, an average of 10.6 days
  If a participant expires during the acute hospitalization, all-cause in-patient mortality will be recorded as described in the electronic medical record including 24 hours after death
Length of acute hospital stay | At the end of the acute hospitalization, an average of 10.6 days
  Number of days of acute hospitalization as recorded by the site staff, will be collected from the electronic medical record after patient's discharge from acute care for all study participants
Discharge disposition | At the end of the acute hospitalization, an average of 10.6 days
  Discharge disposition - The disposition (also called Status) of the patient at time of hospital discharge (i.e., discharged to home, expired, etc.). For each participant, the discharge disposition, will be collected from the electronic medical record on the last day of acute hospitalization
30-day readmission rate | Within 30 days following the last day of acute hospitalization which is an average of 10.6 days
  The number of re-admissions to acute care at this hospital site in the 30 days following discharge will be collected for all participants.

SECONDARY OUTCOMES:
Usability of VR-therapy | Throughout the acute hospitalization, an average of 10.6 days
  Usability of VR-therapy will be assessed at each study session (every 24-72 hours of the hospital stay) through a semi-structured interview conducted immediately after VR-therapy. Usability of VR-therapy will only be assessed in the intervention arm.
Number of participants with VR-therapy related adverse events as assessed by the post-intervention semi-structured interview and research coordinator observations | Throughout the acute hospitalization, an average of 10.6 days
  Participants in the intervention arm will be asked if the VR head mounted display was painful, too heavy, or otherwise uncomfortable. Participants with hearing aids will be asked if they heard buzzing noises during VR-therapy. Participants will be asked if VR-therapy made them feel nervous/anxious, confused/disoriented, nauseous, or any other negative side effect. The research coordinator will observe participant reactions during VR-therapy and record behavior suggesting an unpleasant experience. Participant reactions during VR-therapy will be monitored and the semi-structured interview will be administered immediately after VR-therapy at each session (every 24-72 hours of the hospital stay) for participants in the intervention arm.
In-Hospital Quality of Life Observational Scale | Throughout the acute hospitalization, an average of 10.6 days
  The scale contains 11 items. Total scores range from -22 to 22. Higher scores indicate a higher in-hospital quality of life. This scale is adapted from the Quality of Life in Late-Stage Dementia (QUALID) Scale. Scale will be administered at the beginning of each study session (every 24-72 hours of the hospital stay) for all participants.
Participant Experience and Satisfaction of VR-therapy | Throughout the acute hospitalization, an average of 10.6 days
  Participants in the intervention arm will be asked if they had fun and felt relaxed during VR-therapy. They will be asked open-ended questions about what content they enjoyed most and would like to see in the future. They will be asked if they would like to own VR, recommend VR to a friend, and would like to try VR again. Participant reactions during VR-therapy will be monitored by the research coordinator. Perceived participant enjoyment, relaxation, and engagement will be recorded. Instances of participant vocalizations and reminiscence will be recorded. Participant experience and satisfaction will be assessed at each study session (every 24-72 hours of the hospital stay) for participants in the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lora Appel, PhD, Principal Investigator — OpenLab, University Health Network
Locations (1):
- Michael Garron Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berman MG, Kross E, Krpan KM, Askren MK, Burson A, Deldin PJ, Kaplan S, Sherdell L, Gotlib IH, Jonides J. Interacting with nature improves cognition and affect for individuals with depression. J Affect Disord. 2012 Nov;140(3):300-5. doi: 10.1016/j.jad.2012.03.012. Epub 2012 Mar 31. PMID 22464936
- [Background] Brodaty H, Donkin M. Family caregivers of people with dementia. Dialogues Clin Neurosci. 2009;11(2):217-28. doi: 10.31887/DCNS.2009.11.2/hbrodaty. PMID 19585957
- [Background] Diette GB, Lechtzin N, Haponik E, Devrotes A, Rubin HR. Distraction therapy with nature sights and sounds reduces pain during flexible bronchoscopy: a complementary approach to routine analgesia. Chest. 2003 Mar;123(3):941-8. doi: 10.1378/chest.123.3.941. PMID 12628899
- [Background] Hughes JC, Louw SJ. Electronic tagging of people with dementia who wander. BMJ. 2002 Oct 19;325(7369):847-8. doi: 10.1136/bmj.325.7369.847. No abstract available. PMID 12386013
- [Background] Kaplan R. The Nature of the View from Home: Psychological Benefits. Sage Publications 33(4): 507-542, 2001.
- [Background] Kaplan S. The restorative benefits of nature: toward an integrative framework. Journal of Environmental Psychology 15: 169-182
- [Background] Morita E, Fukuda S, Nagano J, Hamajima N, Yamamoto H, Iwai Y, Nakashima T, Ohira H, Shirakawa T. Psychological effects of forest environments on healthy adults: Shinrin-yoku (forest-air bathing, walking) as a possible method of stress reduction. Public Health. 2007 Jan;121(1):54-63. doi: 10.1016/j.puhe.2006.05.024. Epub 2006 Oct 20. PMID 17055544
- [Background] Park BJ, Tsunetsugu Y, Kasetani T, Kagawa T, Miyazaki Y. The physiological effects of Shinrin-yoku (taking in the forest atmosphere or forest bathing): evidence from field experiments in 24 forests across Japan. Environ Health Prev Med. 2010 Jan;15(1):18-26. doi: 10.1007/s12199-009-0086-9. PMID 19568835
- [Background] Park SH, Mattson RH. Ornamental indoor plants in hospital rooms enhanced health outcomes of patients recovering from surgery. J Altern Complement Med. 2009 Sep;15(9):975-80. doi: 10.1089/acm.2009.0075. PMID 19715461
- [Background] Robinson L, Hutchings D, Corner L, Beyer F, Dickinson H, Vanoli A, Finch T, Hughes J, Ballard C, May C, Bond J. A systematic literature review of the effectiveness of non-pharmacological interventions to prevent wandering in dementia and evaluation of the ethical implications and acceptability of their use. Health Technol Assess. 2006 Aug;10(26):iii, ix-108. doi: 10.3310/hta10260. PMID 16849002
- [Background] Ulrich RS. View through a window may influence recovery from surgery. Science. 1984 Apr 27;224(4647):420-1. doi: 10.1126/science.6143402.
- [Background] Ulrich, RS. Natural Versus Urban Scenes: Some Psychophysiological Effects. Environment and Behavior 13(5): 523-556, 1981.
- [Background] Ulrich RS. Health Benefits of Gardens in Hospitals. Plants for People International Exhibition Floriade 2002.
- [Background] Ulrich RS, Simons RF, Losito BD, Fiorito E, Miles MA, Zelson M. Stress recovery during exposure to natural and urban environments. Journal of Environmental Psychology 11: 201-230, 1991.
- [Background] Weiner MF, Martin-Cook K, Svetlik DA, Saine K, Foster B, Fontaine CS. The quality of life in late-stage dementia (QUALID) scale. J Am Med Dir Assoc. 2000 May-Jun;1(3):114-6. PMID 12818023
- [Derived] Appel L, Appel E, Kisonas E, Lewis-Fung S, Pardini S, Rosenberg J, Appel J, Smith C. Evaluating the Impact of Virtual Reality on the Behavioral and Psychological Symptoms of Dementia and Quality of Life of Inpatients With Dementia in Acute Care: Randomized Controlled Trial (VRCT). J Med Internet Res. 2024 Jan 30;26:e51758. doi: 10.2196/51758. PMID 38289666
- See also: Elderly women with dementia view virtual reality films and provide feedback on their experience. — https://www.youtube.com/watch?v=N3ywcoqR4Co&feature=youtu.be
- See also: The VRx RCT website offered to participants and/or their substitute decision makers to learn more about VR and the study. — https://www.prescribingvr.com/